CLINICAL TRIAL: NCT06243107
Title: The Effectiveness of Tai-Chi in Cancer Patients Improves Fatigue, Mood, Sleep, Quality of Life and Heart Rate Variability
Brief Title: Promoting the Application of Tai Chi to Improve the Fatigue in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201900504B0
Record Dates: First submitted 2023-12-25; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: cancer; Fatigue; negative mood; quality of life; Sleeping quality
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Quasi-experimental research
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai-chi (Experimental): Tai Chi Chuan Intervention: There are 10 styles ,Each movement is performed for 3 minutes, repeated 10 times, totaling 30 minutes per session. participants will engage Tai Chi practice six times a week for eight weeks.
  Interventions: Behavioral: Tai-chi
- control (No Intervention): routine care

INTERVENTIONS:
Behavioral: Tai-chi — Participants will each receive a Tai Chi manual and have access to an instructional audio-visual material via a QR code. The instructional material is tailored specifically for cancer patients. Participants will receive individualized guidance and instructions from the researcher (YH) until they have completed all the executions on the checklist to the required standards.
  Arms: Tai-chi

SUMMARY:
Cancer patients often experience Cancer-Related Fatigue (CRF) due to surgeries, radiation therapy, and/or chemotherapy. CRF does not improve with sleep or rest and not only affects daily activities but can also significantly reduce quality of life. Therefore, finding ways to alleviate fatigue is crucial for cancer patients. Literature indicates that exercise has demonstrated effectiveness in reducing fatigue. Qigong/Tai Chi, based on movement, is a traditional Chinese mind-body practice falling within the range of low to moderate-intensity aerobic exercise. There is no consistent consensus on the effectiveness and frequency of Qigong/Tai Chi for CRF in different cancer patients. Hence, this study aims to investigate through empirical nursing procedures whether "the practice of Qigong/Tai Chi by cancer patients can improve participants' fatigue. Researchers hope that the results of this study can serve as a reference for future clinical applications in alleviating fatigue among cancer patients.

DETAILED DESCRIPTION:
Cancer has consistently ranked as the leading cause of death in Taiwan since 1982. Cancer patients undergo a series of medical treatments, including surgery, radiation therapy, and chemotherapy. Apart from the disease itself, the medical procedures associated with cancer often bring significant physiological, psychological, and emotional stress to the patients. Furthermore, Cancer-Related Fatigue (CRF) is the most common and persistent discomfort experienced by cancer patients. CRF is a prolonged subjective feeling of fatigue or exhaustion that does not improve with sleep or rest. Over 50% of cancer patients report that fatigue reduces participants' physical activity, affects participants ability to perform tasks, and disrupts participants' daily lives, ultimately leading to a diminished quality of life. Among non-pharmacological approaches to managing CRF, exercise has garnered the most research support and demonstrated efficacy. Despite potential limitations on exercise capacity due to the disease, studies have shown that patients, particularly during the initial diagnosis, surgery, or during radiation and chemotherapy, can alleviate CRF and improve participants' overall health through exercise.

Traditional Chinese Exercise and Health Preservation involves using techniques that regulate the mind, breath, and body to promote sufficient qi and blood circulation, unobstructed meridians, and harmonized organ functions. It is a traditional health preservation method aimed at enhancing physical fitness and preventing diseases. Tai Chi, a form of TCEHP, is simple to learn, with minimal space requirements. Through an evidence-based approach and a comprehensive review of two articles, it was found that intervention with Tai Chi for a duration of over 8 weeks, with at least 180 minutes per week, effectively alleviates fatigue in breast cancer and lung cancer patients. It also demonstrated positive effects on fatigue levels in head and neck cancer patients undergoing concurrent chemoradiotherapy (CCRT). Given our institution's diverse cancer patient population, primarily comprising head and neck, breast, and gastrointestinal cancer patients, Researchers plan to proceed with the fourth and fifth steps of the evidence-based practice to apply the evidence to patients and evaluate the care outcomes.

Therefore, the objectives of this study are as follows:

To promote the evidence-based application of Tai Chi for cancer patients to improve fatigue.To promote the evidence-based application of Tai Chi for cancer patients to improve sleep quality.

To promote the evidence-based application of Tai Chi for cancer patients to alleviate anxiety and depression.

To promote the evidence-based application of Tai Chi for cancer patients to enhance quality of life.

To promote the evidence-based application of Tai Chi for cancer patients to assess its impact on heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older;
* Diagnosed with tumors and receiving radiation therapy, chemotherapy, or concurrent chemoradiotherapy.
* Able to communicate and cooperate with the executing team.
* Willing to participate in this study.

Exclusion Criteria:

* Diagnosed with severe internal medical conditions, multiple myeloma, or skeletal metastases.
* Evidence of medical contraindications for exercise.
* Regularly practicing health-preserving exercises or other forms of physical activity.
* Communication barriers, unable to cooperate with the execution of actions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
brief fatigue inventory | At enrollment, during the first week, second week, fourth week, and eighth week.
  Mendoza et al. developed the Brief Fatigue Inventory (BFI) in 1999 to rapidly assess the level of fatigue in cancer patients. This scale comprises nine questions. The first three questions assess the level of fatigue, including current fatigue, typical fatigue over the past 24 hours, and worst fatigue over the past 24 hours. The remaining six questions assess the impact of fatigue on daily life over the past 24 hours, covering general activities, mood, walking ability, daily work (including work outside the home and household chores), interaction with others, and enjoyment of life. Scores range from 0 to 10, where 0 indicates no fatigue, and 10 represents the worst imaginable level of fatigue. The scores for the nine questions are then summed and averaged, with higher scores indicating higher levels of fatigue and a more significant impact on daily life.
  Regenerate

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | t enrollment, during the first week, second week, fourth week, and eighth week
  This scale, developed by Buysse et al. in 1989, is a self-administered questionnaire used to assess the sleep patterns of respondents over the past month. The scale consists of seven monitoring items, including sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each item is rated on a four-point Likert scale. The questionnaire score ranges from 0 to 21 points, with higher scores indicating poorer sleep quality. A PSQI score greater than 5 indicates poor sleep quality. The scale has been translated into Chinese by Wang Runqing. The English version demonstrates a Cronbach's alpha reliability coefficient of .75."
Hospital Anxiety and depression Scale | enrollment, during the first week, second week, fourth week, and eighth week
  This scale, developed by Zigmond and Snaith (1983), is primarily designed to measure anxiety and depression in general clinical populations for assessing the severity of emotional disorders. The Hospital Anxiety and Depression Scale (HADS) utilizes a 4-point scoring system, separate scoring for anxiety and depression, and consists of a total of 14 items, with 7 assessing anxiety and 7 assessing depression. The scores for both domains range from 0 to 21 points. Scores less than 7 indicate the absence of anxiety or depression. Scores between 8 and 10 suggest borderline or suspected cases. Scores equal to or greater than 11 indicate the presence of anxiety or depression. This scale is frequently used in research involving cancer patients. The internal consistency reliability for this scale, measured using Cronbach's alpha, is 0.85 for anxiety and 0.81 for depression."
  Regenerate
FACIT-G quality of life | enrollment, during the first week, second week, fourth week, and eighth week
  "This study utilized the FACIT-G scale for self-reporting and design, although it can also be administered through interviews. The scale is structured around four factors: 'Physical Well-being,' 'Social/Family Well-being,' 'Functional Well-being,' and 'Emotional Well-being.' The scale includes two subscales, 'Emotional Well-being' and 'Social/Family Well-being,' and all subscale items contribute to the total score, which represents the sum of subscale scores. For all FACIT scales and symptom indices, a higher score indicates a better quality of life. The Cronbach's alpha for the entire range is 0.89
Heart rate variability | enrollment, during the first week, second week, fourth week, and eighth week."
  The study utilized a Heart Rate Variability (HRV) monitor (Model: 8Z11, WeGene Corporation, Ministry of Health and Welfare Medical Equipment No. 004896, Taiwan) to measure HRV parameters. This device measures and records electrocardiograms, and calculates heart rate, standard deviation, and mean value using each RR interval. Subsequently, it performs frequency domain analysis to derive HRV parameters, including standard deviation of normal-to-normal intervals, low-frequency power, high-frequency power, and the ratio of low-frequency to high-frequency power.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang MD Hsieh, PHD, Study Director — Chang Gung Medical Foundation
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, No.123,Dinghu Rd.,Guishan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
This study aims to investigate the effects of Tai Chi intervention on fatigue, sleep quality, levels of anxiety and depression, quality of life, and heart rate variability between the Tai Chi group and the control group. The results of the data can be shared.
Supporting Information: Study Protocol
Time Frame: From 2023 to 2025.
Access Criteria: email

REFERENCES:
- [Background] Wayne PM, Lee MS, Novakowski J, Osypiuk K, Ligibel J, Carlson LE, Song R. Tai Chi and Qigong for cancer-related symptoms and quality of life: a systematic review and meta-analysis. J Cancer Surviv. 2018 Apr;12(2):256-267. doi: 10.1007/s11764-017-0665-5. Epub 2017 Dec 8. PMID 29222705
- [Result] Zeng Y, Xie X, Cheng ASK. Qigong or Tai Chi in Cancer Care: an Updated Systematic Review and Meta-analysis. Curr Oncol Rep. 2019 Apr 6;21(6):48. doi: 10.1007/s11912-019-0786-2. PMID 30955106
- [Result] Li W, You F, Wang Q, Shen Y, Wang J, Guo J. Effects of Tai Chi Chuan training on the QoL and psychological well-being in female patients with breast cancer: a systematic review of randomized controlled trials. Front Oncol. 2023 May 1;13:1143674. doi: 10.3389/fonc.2023.1143674. eCollection 2023. PMID 37197428
- [Result] Song S, Yu J, Ruan Y, Liu X, Xiu L, Yue X. Ameliorative effects of Tai Chi on cancer-related fatigue: a meta-analysis of randomized controlled trials. Support Care Cancer. 2018 Jul;26(7):2091-2102. doi: 10.1007/s00520-018-4136-y. Epub 2018 Mar 21. PMID 29564620

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT06243107/Prot_SAP_000.pdf